CLINICAL TRIAL: NCT02889614
Title: Prevalence Assessment and Characterization of Psychological Disorders Associated With Hypobetalipoproteinemia
Acronym: HYPOPSY
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0345
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Hypobetalipoproteinemia
MeSH Terms: conditions — Hypobetalipoproteinemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Hypobetalipoproteinemia diagnosis (LDL-C ≤ 50 mg/dL without hypolipidemic treatment) — LDL-C dosage.

SUMMARY:
Familial hypobetalipoproteinemia (FHBL, OMIM # 1707730) is a genetic disorder heterozygotic of LDL-C metabolism. Clinical manifestation range from asymptomatic patients to metabolic (fatty liver, diabetes) or psychiatric disorders still unrecognized. HYPOPSY research, aims to evaluate prevalence of hypobetalipoproteinemia, and to characterize specific related psychiatric disorders.

DETAILED DESCRIPTION:
Familial hypobetalipoproteinemia (FHBL, OMIM # 1707730) is a genetic disorder heterozygotic of LDL-C metabolism (Low Density Lipoprotein - Cholesterol) whose incidence is measured from 1: 500 to 1: 1000. These heterozygous individuals may be asymptomatic or present some clinical (fatty liver, diabetes) or psychiatric manifestations still unrecognized. Moreover, these individuals have mostly a longevity syndrome and cardiovascular protection. The FHBL is often due to mutations of the APOB (APOlipoprotein B), major component of LDL, VLDL (Very Low Density Lipoprotein) and chylomicrons, and in some cases, loss-of-function mutations of the serine protease PCSK9, endogenous inhibitor of the LDL receptor.

HYPOPSY research, aims to evaluate, in a population with psychiatric disorders, the prevalence of hypobetalipoproteinemia, and to characterize specific related psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in mental Disorders Unit in Nantes University Hospital

Exclusion Criteria:

* Minor patient

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in mental Disorders Unit in Nantes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Frequency of hypobetalipoproteinemia (LDL-C ≤ 50 mg/dL without hypolipidemic treatment) among psychiatric patients managed in Nantes University Hospital | Inclusion.
  Dosage of LDL-C

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided